CLINICAL TRIAL: NCT01352611
Title: Open Label Treatment of Severe Tactile Defensiveness With Intrathecal Baclofen
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1109397
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Tactile Defensiveness; Autistic Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- baclofen, intrathecal (Experimental): A single injection of 50 micrograms of baclofen between the 4th and 5th lumbar vertebrae into the spinal fluid.
  Interventions: Drug: baclofen, intrathecal

INTERVENTIONS:
Drug: baclofen, intrathecal — Patients will undergo a standard intrathecal baclofen trial procedure. This procedure consists of a single injection of 50 micrograms of baclofen between the 4th and 5th lumbar vertebrae into the spinal fluid.
  Other Names: Lioresal, intrathecal.

SUMMARY:
The purpose of this study is to determine if intrathecal administration of baclofen can reduce symptoms of severe tactile defensiveness and autism spectrum disorder.

DETAILED DESCRIPTION:
The purpose of this study is to determine if intrathecal administration of baclofen can reduce symptoms of severe tactile defensiveness and autism spectrum disorder.

Some people with autism spectrum disorder do not like to be touched. This is referred to as tactile defensiveness. Baclofen is a drug approved for treatment of spasticity in patients with conditions such as cerebral palsy, spinal cord injury and traumatic brain injury. Intrathecal means that baclofen is administered by injection into the spinal canal. In this study, each patient will undergo a trial administration of intrathecal baclofen and the effect of intrathecal baclofen on symptoms of tactile defensiveness and autism spectrum disorder will be evaluated.

Each patient will have three visits in connection with the study. First, there will be a screening visit in which the investigators determine if the patient is eligible to participate in the study. To participate, each patient must have autism spectrum disorder, severe tactile defensiveness, and meet other listed criteria. At the second visit, each patient will undergo the intrathecal baclofen trial procedure. The procedure used is the standard procedure to determine if intrathecal baclofen is effective for treatment of spasticity. In this study however, instead of evaluating the effect of intrathecal baclofen on spasticity, the investigators will evaluate the effect of intrathecal baclofen on symptoms of tactile defensiveness and autism spectrum disorder. The trial procedure and evaluation will require about one day. At the third visit, the follow up visit, the investigators will evaluate and discuss the patient's response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of autism prior to study entry
2. Exhibits these specific symptoms of autism:

   * Tactile Defensiveness
   * Increased sensitivity to sensory stimulation
3. Patients must be scored as "Always" for "Reacts emotionally or aggressively to touch" on a modified Short Sensory Profile Questionnaire. Additionally, patients must score "Always" or "Frequently" in the other categories of a modified Short Sensory Profile Questionnaire

Exclusion Criteria:

1. Allergy to baclofen or compounds with similar structure
2. Unable to be evaluated by the chosen efficacy measures
3. Any condition that in the opinion of the principal investigator will place the patient at increased risk of adverse events or preclude completion of the study
4. Concomitant use of any medication that in the opinion of the principal investigator is contraindicated with intrathecal baclofen administration
5. Females of child-bearing potential who have a positive urine pregnancy test at visit 2

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Modified Short Sensory Profile. | Baseline and 2, 4, and 6 hours after administration of intrathecal baclofen
  Changes in tactile defensiveness will be documented on the tactile, movement, and visual/auditory sensitivity sub-scales of a Modified Short Sensory Profile.

SECONDARY OUTCOMES:
Clinical Global Impression of Change in Autism Symptoms | Baseline and 2, 4, and 6 hours after administration of intrathecal baclofen
  Changes in symptoms of autism spectrum disorder from pre-treatment baseline to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Reza S. Farid, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital/University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farid, R.S., Nevel, R. and Murdock, F. Effect of Intrathecal Baclofen on Severe Tactile Defensiveness and Symptoms of Autism Spectrum Disorder. Abstract. International Meeting for Autism Research, Philadelphia, PA. May, 2010.
- See also: Link to Citation — http://imfar.confex.com/imfar/2010/webprogram/Paper5955.html